CLINICAL TRIAL: NCT04821544
Title: Effects of Maternal Stress on Human Milk Composition and Subsequent Infant Outcomes
Brief Title: Maternal Stress on Human Milk and Infant Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: Oregon State University (Other); National Institute of General Medical Sciences (NIGMS) (NIH); Kootenai Health (Other)
Responsible Party: Principal Investigator, Yimin Chen, Assistant Professor, University of Idaho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-024; 5U54GM104944-08 (NIH); P20GM152304 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2021-03-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Depression; Preterm Labor
Keywords: Maternal stress; Mindfulness; Human milk bioactives; Infant metabolome; Maternal transcriptome; Infant transcriptome
MeSH Terms: conditions — Depression, Postpartum; Obstetric Labor, Premature | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control group will receive link to a free 8-week Mindfulness Based Stress Reduction intervention AFTER the 8-weel trial period. This group will also receive placebo gummies that appear the same as the vitamin D gummies.
- Mindfulness-based intervention (with a focus on self-compassion; MBSC) (Experimental): 8-week MBSC intervention with a focus on increasing self-compassion. The MBSC program includes previously developed daily mindfulness practices, guided meditations, routine mindfulness prompts, and four video conference group sessions with a certified mindfulness facilitator.
  Interventions: Behavioral: Mindfulness-based intervention (with a focus on self-compassion; MBSC)
- Vitamin D (Experimental): Vitamin D gummies of 2,000 IU/day for 8 weeks.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Behavioral: Mindfulness-based intervention (with a focus on self-compassion; MBSC) — 8-week MBSC intervention with a focus on increasing self-compassion
  Arms: Mindfulness-based intervention (with a focus on self-compassion; MBSC)
Dietary Supplement: Vitamin D — Vitamin D at 2,000 IU/day for 8 weeks.
  Arms: Vitamin D

SUMMARY:
The overarching purpose of this study is to determine if a modified 8-week mindfulness-based intervention (with a focus on self-compassion; MBSC) or 8 weeks of 2000 IU vitamin D supplementation will reduce stress and increase self-compassion in mothers of preterm infants and beneficially modify the human milk produced, and subsequently improve infant health.

DETAILED DESCRIPTION:
During every two-week period, newly admitted infants (both preterm <37 weeks gestational age and term ≥37 weeks gestational age) at performance site Kootenai Health NICU and term infants from the Palouse region will be block randomized to control (standard of care), mindfulness intervention (modified 8-week mindfulness

-based intervention (with a focus on self-compassion; MBSC), or vitamin D supplementation (8-week 2,000 IU vitamin D3 supplementation) groups. The purpose of the nested cohorts is to minimize the postpartum time difference among cohort mothers. Each nested MBSC cohort will undergo the 8-week MBSC intervention with a focus on increasing self-compassion. The MBSC program includes previously developed daily mindfulness practices, guided meditations, routine mindfulness prompts, and four video conference group sessions with a certified mindfulness facilitator.

Maternal data: The Perceived Stress Scale (PSS) and Self-Compassion Scale-Short Form (SCS-SF) will be given to mothers from both groups pre- and post-intervention, and during the 4th week. Saliva, urine, stool, and human milk samples will be collected at the same time points as above. Additional maternal data include: age, race, height, weight (pre-pregnancy and last weight before delivery), parity, delivery mode, chorioamnionitis, preeclampsia, HELLP (hemolysis, elevated liver enzymes, and low platelet) syndrome, antenatal antibiotics, anti-depressants or other mood-altering/neurochemical medications (current and during pregnancy), diagnosis of depression or other mental illness within the previous 5 years, history of postpartum depression and postpartum psychosis, diabetes, hypertension, heart disease, and any inflammatory or autoimmune diseases.

Infant data: Gestational age, birth weight, ventilation requirement, surgical interventions, patent ductus arteriosus, growth, nutrition prescriptions, saliva, urine and stool samples.

Data collection: All data (not including biosamples) will be collected using REDCap hosted within the UI system.

Sample measurements: Maternal salivary cortisol (marker of stress) and oxytocin (marker of anxiety and "social-closeness") concentrations will be measured using ELISA. Human milk proteins will be identified using mass spectrometry-based proteomics. Following proteomic analyses, targeted proteins will be quantified using ELISA and Western Blot. Both maternal and infant saliva, urine and stool samples will be used for metabolomic and transcriptomic sequencing to identify metabolic and molecular changes, respectively, in both mothers and infants. Infant systemic oxidative stress will be measured through urine F2-isoprostanes concentrations (ELISA), and infant intestinal inflammation will be determined with stool calprotectin concentrations (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Mothers of newborn infants at Kootenai Health NICU and the Palouse region

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Stress - Biomarker Change | Baseline to 4 and 8 weeks
  Salivary cortisol - Change from Baseline cortisol to 4 and 8 weeks
Maternal Stress - Psychometric Measure Change | Baseline to 4 and 8 weeks
  Perceived Stress Scale (PSS) - Change from Baseline PSS to 4 and 8 weeks
  The Perceived Stress Scale (PSS) is validated and the most widely used instrument to measure perception of stress. The PSS includes 14 questions inquiring about feelings and thoughts during the past month expressed through frequency. The PSS will be used pre-intervention, post-intervention (8 weeks), and at the mid-point of the intervention (4 weeks). The scale for each question ranges from 0-4. The PSS measures how often the responder found life to be unpredictable, uncontrollable, and overloaded. Higher score indicates higher perceived stress. The total score ranges between 0-56.
Maternal Self-compassion - Biomarker Change | Baseline to 4 and 8 weeks
  Salivary oxytocin - Change from Baseline oxytocin to 4 and 8 weeks
Maternal Self-compassion - Psychometric Measure Change | Baseline to 4 and 8 weeks
  Self-Compassion Scale-Short Form (SCS-SF) - Change from Baseline SCS-SF to 4 and 8 weeks
  The Self-Compassion Scale-Short Form (SCS-SF)19 is a shortened and highly correlated (r ≥ 0.97) scale (12 items) from the original 26-item SCS. The SCS-SF measures six key components of self-compassion using a scale that ranges from 1-5: self-kindness, self-judgement, common humanity, isolation, mindfulness, and over-identification. Self-compassion is associated with psychological well-being and is therefore often measured alongside stress and anxiety. High score indicates higher self-compassion. The total score ranges between 0-60.

SECONDARY OUTCOMES:
Human Milk Proteins & Peptides Change | Baseline to 4 and 8 weeks
  Protein and peptide profiles will be measured using proteomic & peptidomic analyses to assess human milk protein and peptide changes from baseline to 4 and 8 weeks as a function of maternal changes in stress/self-compassion. These are measured outcomes.
Maternal Metabolomic & Transcriptomic Changes | Baseline to 4 and 8 weeks
  Maternal metabolomic pathways & gene activation changes from baseline to 4 and 8 weeks in response to changes in stress/self-compassion. These are measured outcomes.
Infant Metabolomic & Transcriptomic Changes | Baseline to 4 and 8 weeks
  Infant metabolomic pathways & gene activation changes from baseline to 4 and 8 weeks in response to maternal changes in stress/self-compassion, and human milk protein/peptide profile changes. These are measured outcomes.
Maternal Vitamin D Changes | Baseline to 4 and 8 weeks
  Maternal vitamin D status changes in both serum and human milk from baseline to 4 and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Chen, PhD, Principal Investigator — University of Idaho
Locations (1):
- Kootenai Health, Coeur d'Alene, Idaho, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be available upon request.

DOCUMENTS (1):
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04821544/ICF_000.pdf